CLINICAL TRIAL: NCT02213107
Title: A Phase II Study of Enzalutamide Plus Dutasteride/Finasteride as First Line Treatment for Vulnerable Patients ≥ 65 Years With Systemic Prostate Cancer
Brief Title: Enzalutamide & Dutasteride/Finasteride as 1st Line Treatment for Patients =/> 65 Years Old With Prostate Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Chunkit Fung, Principal Investigator, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53018
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
Keywords: prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Dutasteride; Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enzalutamide and dutasteride or finasteride (Experimental): Use of either 1. Enzalutamide and dutasteride or 2. Enzalutamide and finasteride.
  Interventions: Drug: Enzalutamide and Dutasteride or finasteride

INTERVENTIONS:
Drug: Enzalutamide and Dutasteride or finasteride — Use of either two oral drugs together
  1. Enzalutamide by mouth daily and dutasteride by mouth daily or
  2. Enzalutamide by mouth daily and finasteride by mouth daily

SUMMARY:
Determine the effect of enzalutamide and dutasteride or finasteride on the time to prostatic-specific antigen level increase in patients age 65 or older.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effect of enzalutamide and dutasteride or finasteride on the time to prostatic-specific antigen progression in patients aged 65 or older receiving this combination as first line treatment for systemic prostate cancer.

To determine the safety and toxicities of the study drug combination.

To determine the time to prostatic-specific antigen nadir from the start of study treatment and to evaluate the absolute prostatic-specific antigen nadir as a result of the study drug combination

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features.

Patients with systemic prostate cancer as defined by either a) hormonal naïve metastatic prostate cancer with radiographic evidence of visceral or osseous metastasis or b) biochemical recurrence prostate cancer that fulfills all of the following criteria:

A minimum of three rising prostatic-specific antigen levels with an interval of =/> 1 week between each test, The prostatic-specific antigen (PSA) value at the screening visit should be =/> 2 ng/ml prostatic-specific antigen doubling time ≤ 9 months.

Patients should be 65 years or older. Patients who are deemed "not fit" by comprehensive geriatric assessment or at high risk for side effects as determined by the treating physician. A case report form will be used to document the specifics of why each eligible patient is not considered an ideal candidate.

Serum testosterone level > 1.7 nmol/L (50 ng/dL) at the screening visit (non- castrate).

Patients could have received hormonal therapy as part of definitive treatment for previous localized prostate cancer. However, they should be off any hormonal therapy for greater than six months prior to entry to clinical trial.

Eastern Cooperative Oncology Group performance status of 0 to 2. Able to swallow the study drug and comply with study requirements.

Exclusion Criteria:

Severe concurrent disease or infection that, in the judgment of the investigator, would make the patient inappropriate for enrollment.

Known brain metastases. Brain imaging studies are not required for eligibility if the patient has no neurologic signs or symptoms suggestive of brain metastasis. However, if brain imaging studies are performed, they must be negative for disease.

Patient is receiving treatment for another active malignancy excluding localized cutaneous squamous or basal cell carcinoma.

Prior treatment for systemic prostate cancer. Prior treatment with enzalutamide. Treatment with androgen receptor antagonists (bicalutamide, flutamide, nilutamide,), ketoconazole, abiraterone, finasteride, dutasteride, estrogens, or chemotherapy in an adjuvant setting within 6 months of enrollment (Day 1 visit) or plans to initiate treatment with any of these treatments.

Treatment with therapeutic immunizations for prostate cancer (e.g., PROVENGE®) or plans to initiate treatment with any of these treatments during the study period.

Use of herbal products that may decrease prostatic-specific antigen levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone/prednisolone per day within 4 weeks of enrollment (Day 1 visit) or plans to initiate treatment with any of these treatments during the study.

Radiation therapy within 3 weeks (if single fraction of radiotherapy within 2 weeks) and radioisotope therapy within 8 weeks of enrollment (Day 1 visit).

Participation in a previous clinical trial of an investigational agent that blocks androgen synthesis within six months.

Participation in a previous clinical trial of enzalutamide. Use of an investigational agent within 4 weeks of enrollment (Day 1 visit) or plans to initiate treatment with an investigational agent during the study.

Have used or plan to use from 30 days prior to enrollment (Day 1 visit) through the end of the study the following medications known to lower the seizure threshold or increase or decrease the bioavailability of the drug.

Concomitant use of strong or moderately strong Cytochrome P450 isozyme inducers:

Strong Cytochrome P450 isoenzyme 2C8 inhibitors like gemfibrozil, Strong Cytochrome P450 isoenzyme 2C8 inducers like Rifampin, Strong Cytochrome P450 isoenzyme 3A4 inhibitors like Itraconazole, Aminophylline/theophylline, Atypical antipsychotics (e.g., clozapine, olanzapine, risperidone, ziprasidone), Bupropion, Class IA and Class III antiarrhythmics (e.g., amiodarone, bretylium, disopyramide, ibutilide, procainamide, quinidine, sotalol); Dolasetron, Droperidol, Lithium, Macrolide antibiotics (e.g., erythromycin, clarithromycin); Pethidine, Phenothiazine antipsychotics (e.g., chlorpromazine, mesoridazine, thioridazine); Pimozide, Tricyclic and tetracyclic antidepressants(e.g., amitriptyline, desipramine, doxepin, imipramine, maprotiline, mirtazapine).

History of seizure, including any febrile seizure, loss of consciousness, or transient ischemia attack within 12 months of enrollment (Day 1 visit), or any condition that may predispose to seizure (e.g., prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization).

Clinically significant cardiovascular disease including:

Myocardial infarction within 6 months, Uncontrolled angina within 3 months, Congestive heart failure New York Heart Association class 3 or 4, or patients with history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multigated acquisition scan performed within 3 months results in a left ventricular ejection fraction that is =/> 45%, hypotension (systolic blood pressure < 86 millimeters of mercury [mmHg] or bradycardia with a heart rate < 50 beats per minute, uncontrolled hypertension as indicated by a resting systolic blood pressure of 170 mmHg or diastolic blood pressure > 105 mmHg at the Screening or Study Day 1 visit.

Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer within last 3 months).

Major surgery within 4 weeks prior to enrollment (Day 1 visit). Absolute neutrophil count < 1,500/µL, platelet count < 100,000/µL, and hemoglobin < 5.6 mmol/L (9 g/dL) at the Screening visit; (NOTE: patients may not have received any growth factors or blood transfusions within 7 days of the hematologic laboratory values obtained at the Screening visit).

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chunkit Fung, M.D., Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - University of Rochester, Rochester, New York
  - Medical College of Wisconscin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a single arm study that evaluates the effect of enzalutamide and a 5-alpha reductase inhibitor, with either dutasteride or finasteride. The sample size and power calculations were based on considering subjects using enzalutamide and a 5-alpha reductase inhibitor with either dutasteride or finasteride as a single treatment group. As a result, all analyses for study outcome were performed by including subjects using enzalutamide and a 5-alpha reductase inhibitor as one treatment group.
Groups:
- Enzalutamide and Dutasteride or Finasteride: Use of either 1. Enzalutamide and dutasteride or 2. Enzalutamide and finasteride.
  Enzalutamide and Dutasteride or finasteride: Use of either two oral drugs together
  1. Enzalutamide by mouth daily and dutasteride by mouth daily or
  2. Enzalutamide by mouth daily and finasteride by mouth daily
Period: Overall Study
Arm/Group | Enzalutamide and Dutasteride or Finasteride
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This is a single arm study that evaluates the effect of enzalutamide and a 5-alpha reductase inhibitor, with either dutasteride or finasteride. The sample size and power calculations were based on considering subjects using enzalutamide and a 5-alpha reductase inhibitor with either dutasteride or finasteride as a single treatment group. As a result, baseline analysis population was performed by including subjects using enzalutamide and a 5-alpha reductase inhibitor as one treatment group.
Arm/Group | Enzalutamide and Dutasteride or Finasteride
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 78 [66 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Progression Free Survival
Description: Percentage of participants with progression-free survival at 3 years. PSA disease progression is defined as an increase in the PSA that is >=25% and >=2 ng/ml above the nadir PSA value.
Time Frame: 3 years.
Population: This is a single arm study that evaluates the effect of enzalutamide and a 5-alpha reductase inhibitor, with either dutasteride or finasteride. The sample size and power calculations were based on considering subjects using enzalutamide and a 5-alpha reductase inhibitor with either dutasteride or finasteride as a single treatment group. As a result, primary study outcome analyses were performed by including subjects using enzalutamide and a 5-alpha reductase inhibitor as one treatment group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide and Dutasteride or Finasteride
Number analyzed (Participants) | 43
percentage of participants | 85.3 [70.0 to 93.1]

2. Secondary Outcome: Absolute PSA Response
Description: Lowest PSA value achieved.
Time Frame: up to approximately 8 years
Population: This is a single arm study that evaluates the effect of enzalutamide and a 5-alpha reductase inhibitor, with either dutasteride or finasteride. The sample size and power calculations were based on including subjects using enzalutamide and a 5-alpha reductase inhibitor with either dutasteride or finasteride as one treatment group. The analyses for this outcome included subjects using enzalutamide and a 5-alpha reductase inhibitor as one treatment group. One patient has missing data at 8 years
Measure: Median (Full Range); unit: ng/dl
Arm/Group | Enzalutamide and Dutasteride or Finasteride
Number analyzed (Participants) | 42
ng/dl | 0.02 [0 to 2.75]

3. Secondary Outcome: Time to PSA Nadir
Description: Time (months) to achieve the lowest PSA value compared to baseline PSA level
Time Frame: up to approximately 8 years
Population: This is a single arm study that evaluates the effect of enzalutamide and a 5-alpha reductase inhibitor, with either dutasteride or finasteride. The sample size and power calculations were based on including subjects using enzalutamide and a 5-alpha reductase inhibitor with either dutasteride or finasteride as one treatment group. The analyses for this outcome included subjects using enzalutamide and a 5-alpha reductase inhibitor as one treatment group. One subject has missing data at 8 years
Measure: Median (Full Range); unit: months
Arm/Group | Enzalutamide and Dutasteride or Finasteride
Number analyzed (Participants) | 42
months | 8.05 [1.38 to 78.30]

4. Secondary Outcome: Number of Participants Who Experience a Treatment-related Adverse Events.
Description: Adverse events will be defined according to CTCAE version 4.0.
Time Frame: up to approximately 8 years
Population: This is a single arm study that evaluates the effect of enzalutamide and a 5-alpha reductase inhibitor, with either dutasteride or finasteride. The sample size and power calculations were based on including subjects using enzalutamide and a 5-alpha reductase inhibitor with either dutasteride or finasteride as one treatment group. The analyses for this outcome included subjects using enzalutamide and a 5-alpha reductase inhibitor as one treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide and Dutasteride or Finasteride
Number analyzed (Participants) | 43
Participants | 43

5. Other Pre Specified Outcome: Number of Participants With a Change in Bone Density
Description: Change in bone density at week 103 compared to baseline bone density, measured using DEXA study.
Time Frame: baseline to week 103
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Mean Quality of Life
Description: Change in quality of life score at follow up compared to baseline score, using FACT-P survey. The FACT-P survey is a 39 item questionnaire with a score that ranges from 0-156 with higher scores indicating better quality of life.
Time Frame: baseline to week 61
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Comprehensive Geriatric Assessment Domains
Description: Change in comprehensive geriatric assessment domains at follow up compared to baseline evaluation.
Time Frame: Week 1 to approximately 36 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to approximately 8 years
Description: This is a single arm study that evaluates the effect of enzalutamide and a 5-alpha reductase inhibitor, with either dutasteride or finasteride. The sample size and power calculations were based on including subjects using enzalutamide and a 5-alpha reductase inhibitor with either dutasteride or finasteride as one treatment group. The analyses for adverse events included subjects using enzalutamide and a 5-alpha reductase inhibitor as one treatment group.
Groups:
- Use of Enzalutamide and Dutasteride or Finasteride: Use of either 1. Enzalutamide and dutasteride or 2. Enzalutamide and finasteride.
Arm/Group | Use of Enzalutamide and Dutasteride or Finasteride
All-Cause Mortality (participants affected / at risk) | 5/43
Serious Adverse Events (participants affected / at risk) | 26/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Use of Enzalutamide and Dutasteride or Finasteride (N=43)
Abdominal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Aortic valve disease (Cardiac disorders) | 1
Chest pain, cardiac (Cardiac disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Infection and Infestation, Other (Infections and infestations) | 1
gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Atrial fibrilation (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Dysphasia (Nervous system disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hemorrhage (Blood and lymphatic system disorders) | 1
Lung infection (Infections and infestations) | 1
Lyme disease (Infections and infestations) | 1
Myocardial infarction (Cardiac disorders) | 2
Obstruction (Gastrointestinal disorders) | 1
Presyncope (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 2
Urothelial carcinoma in-situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Covid 19 (Infections and infestations) | 1
constipation (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Use of Enzalutamide and Dutasteride or Finasteride (N=43)
Akathisia (Nervous system disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6
Anemia (Blood and lymphatic system disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 11
Athralgia (Immune system disorders) | 12
Breast pain (Reproductive system and breast disorders) | 5
Constipation (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 14
Dizziness (Nervous system disorders) | 15
Dysgeusia (Nervous system disorders) | 9
Fall (Injury, poisoning and procedural complications) | 15
Fatigue (General disorders) | 38
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Gynecomastia (Reproductive system and breast disorders) | 31
Hot flashes (Vascular disorders) | 18
Hypertension (Vascular disorders) | 17
Memory impairment (Nervous system disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Nausea (Gastrointestinal disorders) | 11
Osteoporosis (Musculoskeletal and connective tissue disorders) | 8
Paresthesia (Nervous system disorders) | 9
Weight loss (Investigations) | 5
Abdominal Pain (Gastrointestinal disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 11
AST increased (Investigations) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 9
Blood and Lymphatic Disorders, Other (Blood and lymphatic system disorders) | 4
Blurred Vision (Eye disorders) | 4
Cardiac disorder, other (Cardiac disorders) | 3
Cataract (Eye disorders) | 4
Chest pain, cardiac (Cardiac disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Creatinine increase (Investigations) | 8
Cystitis noninfective (Renal and urinary disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16
Edema of limbs (General disorders) | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Erectile dysfunction (Reproductive system and breast disorders) | 3
Eye disorders, Other (Eye disorders) | 7
Floaters (Eye disorders) | 3
Fracture (Injury, poisoning and procedural complications) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders, other (Gastrointestinal disorders) | 6
General disorders (General disorders) | 6
Headache (Nervous system disorders) | 7
Hearing impaired (Ear and labyrinth disorders) | 3
Hematuria (Renal and urinary disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 6
Infection and Infestation, Other (Infections and infestations) | 4
Injury, poisoning, or procedural complications, other (Injury, poisoning and procedural complications) | 4
Insomnia (Psychiatric disorders) | 6
Lymphocyte Count Decreased (Investigations) | 5
Musculoskeletal and connective tissue disorder, other (Musculoskeletal and connective tissue disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Neoplasms benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Neutrophil count decreased (Investigations) | 3
Non-cardiac chest pain (General disorders) | 9
Pain (General disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Peripheral sensory neuropathy (Nervous system disorders) | 4
Psychiatric disorder, other (Psychiatric disorders) | 3
Rash, maculo-papular (Skin and subcutaneous tissue disorders) | 7
Renal and urinary disorder (Renal and urinary disorders) | 5
Reproductive system and breast disorders, others (Reproductive system and breast disorders) | 4
Respiratory, thoracic, and mediastinal disorders, other (Respiratory, thoracic and mediastinal disorders) | 6
Other Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 9
Upper respiratory infection (Infections and infestations) | 6
Urinary frequency (Renal and urinary disorders) | 6
Urinary incontinence (Renal and urinary disorders) | 8
Urinary tract infection (Infections and infestations) | 4
Urinary urgency (Renal and urinary disorders) | 4
Weight gain (Investigations) | 5
White blood cell decreased (Investigations) | 4
Aortic valve disease (Cardiac disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT02213107/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT02213107/ICF_001.pdf